CLINICAL TRIAL: NCT03410368
Title: A Randomized, Controlled, Open-label, Single Center, Phase II Study to Evaluate the Efficacy and Safety of NK Cell-based Immunotherapy as Maintenance Therapy for Patients With Small-cell Lung Cancer After First-line Chemotherapy.
Brief Title: NK Cell-based Immunotherapy as Maintenance Therapy for Small-Cell Lung Cancer.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: jiuwei cui (Other)
Responsible Party: Sponsor-Investigator, jiuwei cui, chief, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FHJLU-001
Record Dates: First submitted 2017-12-28; First posted 2018-01-25 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Small Cell Lung Cancer
Keywords: maintenance therapy; immunotherapy; adoptive cell transfer; natural killer cell
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Intervention Model Description: Patients with small-cell lung cancer receive autologous NK cells adoptive cancer immunotherapy as a maintenance therapy in the presence of stable disease (SD), partial remission (PR) or complete remission (CR) after the first-line chemotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- autologous natural killer cells (Experimental): Infusion of 1-2×10^9 NK cells every 14 days in the absence of progression or unacceptable toxicity until the 6 courses of treatment.
  Interventions: Biological: NK cells
- routine follow-up (No Intervention): According to present guideline, no special treatment is advised for patients with SCLC after first-line therapy.They will be followed-up regularly.

INTERVENTIONS:
Biological: NK cells — Autologous peripheral blood mononuclear cells (PBMCs) are collected by apheresis on D0, then induced into NK cells and infused into the patients 14 days later (D14) as the initial transfusion. There are 3 consecutive transfusion days (D14-D16). The second course of PBMCs collection started D14 before infusion. A total of 6 courses will be completed unless progression or unacceptable adverse events.
  Arms: autologous natural killer cells

SUMMARY:
Natural killer (NK) cells can kill a broad array of tumor cells in a non-major histocompatibility complex(MHC)-restricted manner. Adoptive transfer of NK may prolong the survival of patients with cancer. This study evaluates the efficacy and safety of NK cell-based immunotherapy for small-cell lung cancer (SCLC) after first-line chemotherapy. Half of the participants will receive autologous adoptive transfer of NK cells after the response from first-line chemotherapy, while the other half will be followed up in routine clinal practice.

DETAILED DESCRIPTION:
The small-cell lung cancer (SCLC) is very sensitive to the standard-of-care first-line chemotherapy and/or radiotherapy, but it will ultimately progress or relapse and develop early resistance to conventional treatments. No effective maintenance therapy except for wath and wait after first-line therapy at present.

NK cells constitute the major component of the innate immune system and kill tumor cells in a non-MHC-restricted manner. In our previous pilot study and other reports, adoptive transfer of autologous NK cells expanded ex vivo was very well tolerant and effective.

There is no prospective trial on the maintenance therapy of SCLC after first-line chemotherapy based on autologous NK cells. The purpose of this phase II clinical research is to evaluate the efficacy and safety of autologous NK cells as the maintenance therapy after the first-line treatment, comparing with conventional observation group.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed small cell lung cancer.
* Having completed first-line therapy in the presence of stable disease (SD), partial remission (PR) or complete remission (CR) status.
* Age ≥18 years.
* Karnofsky Performance Status (KPS) ≥80.
* Important organs:cardiac ejection fraction >50%; Pulse Oxygen Saturation(SpO2) >90%; creatinine (Cr) ≤ 2.5 times the normal range; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 times the normal range, total bilirubin (TBIL)≤2.0mg/dl (34.2umol/L);Hgb≥60g/L.
* Without contraindication of apheresis and cell isolation.
* Patients and their families having the willingness to participate in clinical trial with signed written informed consent.

Exclusion Criteria:

* Patient having an active rheumatic immunologic disease.
* Uncontrolled bacterial, fungal or viral infection.
* human immunodeficiency virus(HIV), hepatitis B virus infection(HBV), hepatitis C virus(HCV) infection.
* History of organ transplantation and hemopoietic stem cell transplantation.
* Pregnant or lactating women.
* Patients using immunosuppressive agents within the first 3 months of the study or received glucocorticoid systemic therapy within a week prior to entry into the study.
* Patients receiving other immunotherapy after diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | 20 months
  Progression-free survival is defined as the time from randomization to first observation of progression or date of death (from any cause). Progression will be evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. Patients who do not progress or not die will be censored on the date of their last tumor assessment, i.e. on the last date that we really know that the patient is considered as "progression-free".

SECONDARY OUTCOMES:
Overall survival(OS) | 20 months
  Overall survival, defined as the time from randomization until death due to any cause. For patients who do not die, time to death will be censored at the time of the last contact.
Evaluate the change of the quality of life for all patients | 20 months
  Patients' quality-of-life will be assessed by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 and European Organization for Research and Treatment of Cancer Quality of Life Questionnaire LC-13 at baseline and after every two courses of adoptive cellular transfer in study group or every visit in control group.

CONTACTS AND LOCATIONS:
Overall Officials: jiuwei cui, PhD, Principal Investigator — the Cancer Center of First Hospital of Jilin University
Locations (1):
- the First Hospital of Jilin University, Ch’ang-ch’un, Jilin, China

IPD SHARING:
Plan to Share IPD: No